CLINICAL TRIAL: NCT03290651
Title: Re-setting the Breast Microbiome to Lower Inflammation and Risk of Cancer.
Brief Title: Probiotics and Breast Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Muriel Brackstone, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 110181
Record Dates: First submitted 2017-09-14; First posted 2017-09-25 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Intervention Model Description: Double blind randomized, placebo-controlled pilot trial.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Natural Health Product - RepHresh Pro-B (Experimental): One capsule contains 2.5 billion CFU of Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14.
  Interventions: Dietary Supplement: Probiotic Natural Health Product - RepHresh Pro-B
- Placebo (Placebo Comparator): Placebo. It is the same composition as the active capsule, without the bacteria.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Natural Health Product - RepHresh Pro-B — Participants will take the probiotic or placebo daily for 90 days.
  Arms: Probiotic Natural Health Product - RepHresh Pro-B
Dietary Supplement: Placebo — Participants will take the probiotic or placebo daily for 90 days.
  Arms: Placebo

SUMMARY:
Breast cancer remains a major killer of women and despite major advances in care, the role of 'environmental factors' in the disease remain to be well understood. The investigators have shown that one such factor is the bacteria that inhabit the breast tissue. These bacteria do not cause infections per se, but can produce low amounts of substances known to be able to induce cancer. The investigators have found that the bacteria in the breasts of women with cancer are very different from those found in the breast tissue of healthy women. The investigators would like to test their theory that taking probiotic lactobacilli by mouth can lead to these organisms reaching the breast tissue and help to displace the harmful bacteria and reduce inflammation which has close links to cancer.

DETAILED DESCRIPTION:
Certain bacteria, particularly Gram negatives, are major causes of inflammation. In fact, the lipopolysaccharides from these bacteria are used in vast numbers of studies to induce inflammation and study disease. Many cancers are the result of inflammatory processes. Breast cancer is a major cause of illness and death in women and inflammatory processes are one of the foci of investigation; however, not yet from the stand point that bacteria in the breast may be the instigators of cancer development. The investigators were the first in the world to describe the breast microbiota and show that the bacterial profiles are more pathogenic in women with cancer than in tissues of healthy controls. This work has been validated by others. Although this does not prove a cause-and-effect link with breast cancer, such linkages have been shown in stomach and colon cancers. If researchers assume there is a link, then how can the inflammatory microbiota be re-set to one that is somehow beneficial and able to reduce inflammation and potential cancer induction?

The concept of probiotics emerged from the quest to reset the disrupted microbiota of the gut and upper respiratory tract. This investigational group has led the world in doing the same in the urogenital tract of women.

The researchers would like to test their theory that taking probiotic lactobacilli by mouth can lead to these organisms reaching the breast tissue and helping displace the harmful bacteria and reducing inflammation. A study in Spain has shown that oral intake of probiotic lactobacilli can not only cure mastitis, but lead to the lactobacilli reaching the milk glands. Women who breast feed for more than six months (and thereby pass along lactic acid bacteria to the infant from the breast milk) have a reduced risk of breast cancer.

The investigators hypothesize that the breast microbiome of women at risk of cancer has the same profile as women with cancer and that oral administration of probiotic lactobacilli can reset this to one found in healthy women. They also hypothesize the breast tissue of these at-risk patients is contaminated by environmental toxins.

The project plan is to test the concept of re-setting the breast tissue microbiota in women at risk of cancer, to one more aligned with health.

Samples will be tested for relative bacterial abundance to determine any shift in bacterial breast tissue composition by next-generation sequencing and bioinformatics. Samples will also be tested for inflammatory markers using Luminex technology, and for mercury, arsenic and pesticides using LC-MS as described in previous studies.

Twenty women at high-risk for breast cancer (See Inclusion Criteria) will be randomized (10 each) to receive either probiotic or placebo, once a day for 90 days. This capsule is approved in Canada and widely available and contains 2.5 billion CFU viable bacterial cells of each of the following strains: Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14. Both active capsules and placebo will be provided by the manufacturer Chr Hansen (Denmark). Samples will be collected at t=0 (enrollment), t=1 (end of 90 days) and t=2(30 days post-treatment).

Twenty women will act as healthy controls (See Inclusion Criteria) and will be randomized (10 each) as described above for the high-risk group.

At each time point, samples collected will include:

* Breast skin swab - a cotton tipped swab with be moistened with sterile water and the passed over the skin on the breast 10 times.
* Needle aspirate - a 22-gauge needle into the breast tissue with repeated passage under suction until aspirate material is identified in the needle hub. This material would then be placed in normal saline.
* Nipple aspirate - the participant will be asked to massage their breast from chest wall to nipple for several minutes as needed. Using a hand-held modified breast pump placed over the nipple, nipple aspirate fluid will be drawn out and into a capillary tube.
* Blood draw - one 6mL EDTA plasma tube using standard phlebotomy procedures. Samples will be analyzed for relative bacterial abundance (next-generation sequencing), inflammatory markers (Luminex technology).
* Urine - 100mL sample that will be tested for heavy metals and pesticides using LC-MS.

ELIGIBILITY:
Inclusion Criteria:

* Women at high risk of developing breast cancer who have never had breast cancer (≥ 25% lifetime risk and/or BRCA1 or BRCA2 positive) will be included in the high risk group, while female family members of cancer patients or friends of patients, as well as patients to the breast clinic who are seen for other reasons not related to cancer will be offered participation in the control group.

Exclusion Criteria:

* Exclusion criteria include: immunosuppression (ongoing high dose steroids, immunosuppressive condition such as HIV), personal history of breast cancer, patients declining needle aspiration biopsy or probiotic/placebo treatment, ongoing daily oral probiotic treatment at time of diagnosis. Patients on chronic or recent (within 2 weeks) antibiotic therapy will also be excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in breast microbiota | 90 days post collection period
  The diversity of the breast microbiota analysed using next-generation sequencing.

SECONDARY OUTCOMES:
Testing of inflammatory markers and pollutants | 90 days post collection period
  Blood samples will be testing by luminex for inflammatory cytokine/chemokine markers.
Testing for environmental pollutants - heavy metals. | 90 days post collection period
  Urine and blood will be tested for heavy metals using LC-MS.
Testing for environmental pollutants - pesticides. | 90 days post collection period
  Urine and blood will be tested for pesticides using LC-MS.

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Reid, Ph.D., Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Muriel Brackstone, M.D., Principal Investigator — St. Joseph's Health Care London
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arroyo R, Martin V, Maldonado A, Jimenez E, Fernandez L, Rodriguez JM. Treatment of infectious mastitis during lactation: antibiotics versus oral administration of Lactobacilli isolated from breast milk. Clin Infect Dis. 2010 Jun 15;50(12):1551-8. doi: 10.1086/652763. PMID 20455694
- [Background] Urbaniak C, Cummins J, Brackstone M, Macklaim JM, Gloor GB, Baban CK, Scott L, O'Hanlon DM, Burton JP, Francis KP, Tangney M, Reid G. Microbiota of human breast tissue. Appl Environ Microbiol. 2014 May;80(10):3007-14. doi: 10.1128/AEM.00242-14. Epub 2014 Mar 7. PMID 24610844
- [Background] Urbaniak C, Gloor GB, Brackstone M, Scott L, Tangney M, Reid G. The Microbiota of Breast Tissue and Its Association with Breast Cancer. Appl Environ Microbiol. 2016 Jul 29;82(16):5039-48. doi: 10.1128/AEM.01235-16. Print 2016 Aug 15. PMID 27342554
- [Background] Hieken TJ, Chen J, Hoskin TL, Walther-Antonio M, Johnson S, Ramaker S, Xiao J, Radisky DC, Knutson KL, Kalari KR, Yao JZ, Baddour LM, Chia N, Degnim AC. The Microbiome of Aseptically Collected Human Breast Tissue in Benign and Malignant Disease. Sci Rep. 2016 Aug 3;6:30751. doi: 10.1038/srep30751. PMID 27485780
- [Background] Chan AA, Bashir M, Rivas MN, Duvall K, Sieling PA, Pieber TR, Vaishampayan PA, Love SM, Lee DJ. Characterization of the microbiome of nipple aspirate fluid of breast cancer survivors. Sci Rep. 2016 Jun 21;6:28061. doi: 10.1038/srep28061. PMID 27324944
- [Background] Zackular JP, Baxter NT, Iverson KD, Sadler WD, Petrosino JF, Chen GY, Schloss PD. The gut microbiome modulates colon tumorigenesis. mBio. 2013 Nov 5;4(6):e00692-13. doi: 10.1128/mBio.00692-13. PMID 24194538
- [Background] Mira-Pascual L, Cabrera-Rubio R, Ocon S, Costales P, Parra A, Suarez A, Moris F, Rodrigo L, Mira A, Collado MC. Microbial mucosal colonic shifts associated with the development of colorectal cancer reveal the presence of different bacterial and archaeal biomarkers. J Gastroenterol. 2015 Feb;50(2):167-79. doi: 10.1007/s00535-014-0963-x. Epub 2014 May 9. PMID 24811328
- [Background] Sitas F. Twenty five years since the first prospective study by Forman et al. (1991) on Helicobacter pylori and stomach cancer risk. Cancer Epidemiol. 2016 Apr;41:159-64. doi: 10.1016/j.canep.2016.02.002. Epub 2016 Feb 26. PMID 26922171
- [Background] Macklaim JM, Clemente JC, Knight R, Gloor GB, Reid G. Changes in vaginal microbiota following antimicrobial and probiotic therapy. Microb Ecol Health Dis. 2015 Aug 14;26:27799. doi: 10.3402/mehd.v26.27799. eCollection 2015. PMID 26282697
- [Background] Bisanz JE, Enos MK, Mwanga JR, Changalucha J, Burton JP, Gloor GB, Reid G. Randomized open-label pilot study of the influence of probiotics and the gut microbiome on toxic metal levels in Tanzanian pregnant women and school children. mBio. 2014 Oct 7;5(5):e01580-14. doi: 10.1128/mBio.01580-14. PMID 25293764
- [Background] Bisanz JE, Seney S, McMillan A, Vongsa R, Koenig D, Wong L, Dvoracek B, Gloor GB, Sumarah M, Ford B, Herman D, Burton JP, Reid G. A systems biology approach investigating the effect of probiotics on the vaginal microbiome and host responses in a double blind, placebo-controlled clinical trial of post-menopausal women. PLoS One. 2014 Aug 15;9(8):e104511. doi: 10.1371/journal.pone.0104511. eCollection 2014. PMID 25127240